CLINICAL TRIAL: NCT01324609
Title: Detection of Choroidal Nevus Cells in Vitrectomy Fluid
Status: Terminated | Type: Observational
Why Stopped: Could not recruit enough patients
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Darius M. Moshfeghi, Principle Investigator, Stanford University
Other Study IDs: SU-03242011-7564; IRB-18580
Record Dates: First submitted 2011-03-25; First posted 2011-03-29 (Estimated); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Nevus
Keywords: choroidal nevus; vitrectomy
MeSH Terms: conditions — Nevus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to determine if the investigators can detect the presence of choroidal nevi cells in the vitreous fluid of humans, as this may improve the diagnosis and classification of choroidal nevi and melanomas in the future.

DETAILED DESCRIPTION:
Approximately 7% of the population has a choroidal nevus, or "freckle," in the back of the eye. Like a nevus on the skin, there is potential for malignant change to a melanoma. Dermatologists have the ability to quickly and easily biopsy suspicious skin lesions while ophthalmologists currently have no way of determining the malignant potential of choroidal nevi other than a fine needle aspiration (which is invasive and has the potential complications of bleeding and retinal detachment). This study's sole aim is to see if choroidal nevi cells are present in the inside fluid of the eye. The investigators plan to analyze the fluid of the eye, which is routinely removed during retina surgery, to detect any nevus cells. If the investigators are able to detect these cells, then future studies may allow us to better classify choroidal nevi for potential malignant change.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a choroidal nevus who are undergoing routine vitrectomy surgery for another indication (such as epiretinal membrane or macular hole repair).

Exclusion Criteria:

* Patients without a choroidal nevus
* Children under the age of 18
* Pregnant and nursing females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a choroidal nevus who are undergoing routine vitrectomy surgery for another indication.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2010-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Positive identification of nevus cells in eye fluid | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Darius M. Moshfeghi, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States